CLINICAL TRIAL: NCT06693206
Title: Investigation of Burnout, Musculoskeletal System, Physical Performance and Perception of Exercise Benefit / Obstacle and Aerobic Capacity in Nurses
Brief Title: Investigation of Burnout, Musculoskeletal System and Aerobic Capacity in Nurses
Status: Not yet recruiting | Type: Observational
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Songül Bağlan Yentür, Head of Physiotherapy and Rehabilitation Department, Firat University
Other Study IDs: 2024/13-05
Record Dates: First submitted 2024-11-14; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Aerobic Capacity
Keywords: nurse; aerobic capacity; burnout
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Nurse group: Nurses will be evaluated in terms of burnout, aerobic capacity and musculoskeletal pain.
  Interventions: Other: Evaluation of aerobic capacity

INTERVENTIONS:
Other: Evaluation of aerobic capacity — A stepwise protocol will be used in which the load increases gradually with the bicycle ergometer. In these protocols, the load increases continuously in small amounts throughout the exercise.

SUMMARY:
The aim of our study was to evaluate the relationship of aerobic capacity with burnout status, musculoskeletal system, physical performance and exercise benefit/obstacle perception in nurses, who have an important place in the health profession group, and to bring the results to the literature. Demographic information will be obtained from the participants who volunteered to participate in the study. Burnout, musculoskeletal pain and physical performance will be evaluated with relevant scales and aerobic capacity will be measured with a bicycle ergometer.

DETAILED DESCRIPTION:
In the literature, there are studies on the general effects of aerobic exercises on the cardiovascular system, musculoskeletal system, endocrine system, nervous system and psychosocial status. However, despite the benefits of aerobic exercises and the physiological and psychological importance of high aerobic capacity, there are no studies in the literature that examine the factors associated with the aerobic capacity of nurses. These factors affect the professional life of nursesThe aim of our study was to evaluate the relationship of aerobic capacity with burnout status, musculoskeletal system, physical performance and exercise benefit/obstacle perception in nurses, who have an important place in the health profession group, and to bring the results to the literature. Demographic information will be obtained from the participants who volunteered to participate in the study. Burnout, musculoskeletal pain and physical performance will be evaluated with relevant scales and aerobic capacity will be measured with a bicycle ergometer.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* At least 1 year of experience
* Nurses not working in the academic field

Exclusion Criteria:

* Pregnancy
* Malignancy
* Nurses with lower extremity problems

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include 30 female nurses who work in Fırat University Hospital on normal shift and do not have any chronic disease.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-11-10 (Estimated); Primary Completion 2024-12-10 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Aerobic capacity assessment | up to 30 minutes
  A stepwise protocol will be used in which the load increases gradually with the bicycle ergometer. In these protocols, the load increases continuously in small amounts throughout the exercise.

SECONDARY OUTCOMES:
Burnout assessment | up to 30 minutes
  Maslach Burnout Inventory, which was developed by Christina Maslach and Susan Jackson (1986) and Turkish adaptation and validity-reliability study was conducted by Ergin (1992), will be completed. The 7-point Likert-type scale, which consists of 22 items in total and consists of 'Never- Few Times a Year- Few Times a Month- Once a Month- Few Times a Week- Once a Week- Every Day' options in its original form, was reduced to five options in the adaptation study conducted by Ergin (1992) on the grounds that it was not suitable for Turkish culture.
Musculoskeletal evaluation | up to 30 minutes
  n 1987, the Nordic Musculoskeletal Questionnaire developed by Kuorinka to measure musculoskeletal pain will be completed. The body is divided into 9 regions: neck, shoulder, back, elbow, hand/wrist, waist, hip/thigh, knee, foot/ankle. It is assessed whether there is a problem in these areas and if so, how long it has been going on

CONTACTS AND LOCATIONS:
Overall Officials: Songul Baglan Yentur, Principal Investigator — Firat University

IPD SHARING:
Plan to Share IPD: No